CLINICAL TRIAL: NCT02840084
Title: A Study on the Safety and Effectiveness of the Aspen™ Ultrasound System and Aspen Rehabilitation Technique in the Treatment of Capsular Contracture Baker Grade III
Brief Title: Aspen™ Ultrasound System and Aspen Rehabilitation Technique in the Treatment of Capsular Contracture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: adverse event
Sponsor: Nina Naidu (Individual)
Responsible Party: Sponsor-Investigator, Nina Naidu, Plastic & Reconstructive Surgeon, Naidu, Nina S., M.D.
Organization: Naidu, Nina S., M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G160087
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Capsular Contracture of Breast, Grade III
Keywords: breast implant capsular contracture
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Patients (Experimental): In stage I, 10 women aged 22 years or older who have received silicone or saline breast implants for subglandular or submuscular breast augmentation, and who subsequently developed Baker Grade III capsular contracture, will be invited to participate. In Stage II, the study group will be expanded to include an additional 50 patients who have received saline or silicone gel implants, placed in either the subglandular or submuscular position, with Grade III capsular contracture of the breast. The intervention will be treatment with the Aspen(TM) Ultrasound System.
  Interventions: Device: Aspen(TM) Ultrasound System

INTERVENTIONS:
Device: Aspen(TM) Ultrasound System — Two transducers per breast are applied. There will be 10 30 minute sessions, with 2 sessions per week for five weeks. The transducers will be placed on the medial and lateral positions of the affected breast, and then rotated to the superior and inferior aspects, and finally directly over the nipple-areolar complex. Following treatment, the affected breast will be massaged and bandaged per the Aspen Rehabilitation protocol, and the patient will be provided with home exercises as part of the Aspen Rehabilitation Technique.
  The treated breast(s) will be examined both prior to and immediately following each treatment session. To evaluate safety, any adverse events such as swelling, redness, or pain will be assessed. To determine efficacy, any change in the Baker Grade level will be assessed by physical examination. The breasts will be photographed prior to treatment at each visit to assist in evaluation of any visible change in the breasts.

SUMMARY:
Purpose: The purpose of this investigation is to test the safety and effectiveness of the Aspen System™ and Aspen Rehabilitation Technique. The device is intended for the therapeutic treatment of capsular contracture of the breast in conjunction with the Aspen Rehabilitation Technique. The hypothesis of the proposed study is that external ultrasound with the Aspen System™ device in conjunction with the Aspen Rehabilitation Technique is safe and effective in the reduction by at least one level of Baker Grade III capsular contracture in cosmetic breast augmentation patients, maintained at one year from the final treatment. Potential benefits of the study to subjects include improvement in the grade of capsular contracture of the breast without surgical treatment. The investigation is planned to last 12 months.

DETAILED DESCRIPTION:
Protocol:

Objectives: Two stages are proposed for this study. In Stage I, the objective is to demonstrate the safety of the Aspen System™ and Aspen Rehabilitation Technique in the treatment of Baker Grade III capsular contracture of the breast following subglandular or submuscular placement of saline or silicone implants for cosmetic breast augmentation. The endpoint will be the determination of safety as defined by no adverse events, including implant rupture. Following review of interim data and approval by the FDA, Stage II will commence. In Stage II, the objective will be to demonstrate safety and efficacy of the Aspen System™ and Aspen Rehabilitation Technique in the treatment of Baker Grade III capsular contracture of the breast following subglandular or submuscular placement of saline or silicone implants for cosmetic breast augmentation. The endpoint will be the documentation of efficacy as demonstrated by the reduction of at least one Baker Grade following treatment with the Aspen™ System and Aspen Rehabilitation Technique.

Description: This is a prospective, non-randomized trial.

Conduct: The trial will be conducted as follows:

Study Subjects: Patients will be recruited from the investigator's private practice and the local community. In stage I, 10 women aged 22 years or older who have received saline or silicone breast implants for subglandular or submuscular breast augmentation, and who subsequently developed Baker Grade III capsular contracture, will be invited to participate. Upon completion of the first stage of this study, the data will be submitted to the FDA for review. The second stage of the study will not commence until approval has been obtained by the FDA. At this time, for the second stage of the study, the study group will be expanded to include an additional 50 patients who have received saline or silicone gel implants, placed in either the subglandular or submuscular position, with Grade III capsular contracture of the breast.

ELIGIBILITY:
Inclusion Criteria:

Stage I:

* Age 22 years or greater,
* Cosmetic breast augmentation,
* Baker Grade III capsular contracture, subglandular implant position, saline implants.

Stage II:

* Age 22 years or greater,
* Cosmetic breast augmentation,
* Baker Grade III capsular contracture, subglandular or submuscular implant position, saline or silicone gel implants.

Exclusion Criteria:

* History of breast cancer,
* prior radiation therapy to chest wall,
* ruptured breast implant,
* calcification of capsules seen on any imaging study,
* implants > 15 years old,
* prior treatment for capsular contracture in past 12 months (open capsulectomy, open capsulotomy, implant exchange, implant plane change, placement of acellular dermal matrix, explantation, closed capsulotomy, or oral medication),
* metal implants,
* pacemakers,
* defibrillators,
* history of epilepsy,
* history of bleeding, and undiagnosed pain syndromes,
* pregnancy,
* currently lactating,
* acute and sub-acute thrombosis and thrombophlebitis,
* potentially malignant tumors,
* benign tumors,
* malignancy,
* third-degree musculotendinous lesions,
* multiple sclerosis,
* osteomyelitis,
* cardiac arrhythmias,
* acute sepsis of tissue or bone,
* arteriosclerosis,
* hemophilia, and
* sensory nerve damage.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Safety (defined by no adverse events, including implant rupture, skin burns) of the Aspen™ Ultrasound System and Aspen Rehabilitation Technique in the Treatment of Capsular Contracture Baker Grade III | 12 months
  The determination of safety as defined by no adverse events, including implant rupture, skin burns,
Efficacy (reduction of at least one Baker Grade following treatment) of the Aspen™ Ultrasound System and Aspen Rehabilitation Technique in the Treatment of Capsular Contracture Baker Grade III | 12 months
  The documentation of efficacy as demonstrated by the reduction of at least one Baker Grade following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Naidu, MD, Principal Investigator — surgeon
Locations (1):
- Nina S. Naidu, MD PC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Non-identified data may be made available to the FDA if requested.